CLINICAL TRIAL: NCT05574348
Title: Effect of Osteopathic Protocol in 2 Sessions (PO2S) for Patients With Non-specific Spine: a Randomized Cross-over Clinical Trial
Brief Title: Evaluation of Osteopathic Protocol on Rachialgia
Acronym: PO2S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cabinet d'ostéopathie Michel Boeuf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PO2S
Record Dates: First submitted 2022-10-04; First posted 2022-10-10 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Spine Injuries and Disorders
Keywords: Osteopathic; Pain; Spine
MeSH Terms: conditions — Disease; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PO2S - Control (Experimental): This arm will start with PO2S, followed by Control. The PO2S consists of two sessions of 30 minutes each, one week apart, composed of normalizations of joint, muscular, ligament and visceral dysfunctions .
  Control is a treatment in 2 sessions that is like PO2S but is not an active osteopathic treatment. A light touch will be made for fictitious normalizations.
  Interventions: Other: Osteopathic Protocol in 2 Sessions (PO2S)
- Control - PO2 (Experimental): This arm will start with Control, followed by PO2S. The PO2S consists of two sessions of 30 minutes each, one week apart, composed of normalizations of joint, muscular, ligament and visceral dysfunctions .
  Control is a treatment in 2 sessions that is like PO2S but is not an active osteopathic treatment. A light touch will be made for fictitious normalizations.
  Interventions: Other: Osteopathic Protocol in 2 Sessions (PO2S)

INTERVENTIONS:
Other: Osteopathic Protocol in 2 Sessions (PO2S) — PO2S works on the principle that there is a concordance between the author's Preferential Torsion Pattern (PTP) and the rotatory direction of osteopathic dysfunctions.
  The PO2S consists of two sessions of 30 minutes each, one week apart. A 13-item clinical examination is performed at the first session. It focuses on caused pain tests, and classifies patients in left or right PTP. During the first session 14 normalizations of joint, muscular, ligament and visceral dysfunctions are performed systematically. During the second session 10 normalizations of joint, muscular, ligament and visceral dysfunctions are performed .
  PO2S is an innovative osteopathic protocol for back pain.

SUMMARY:
Rachialgia are among the most common reasons for consultation with the general practitioner in Europe. Most of the guidelines recommend spinal manipulation.

This study attempts to propose a solution with 2 parts: tests of induced pain that have a greater sensitivity than palpatory tests of movements and a comprehensive musculoskeletal treatment protocol.

The aim of this study is to evaluate the Osteopathic Protocol in 2 sessions (PO2).

DETAILED DESCRIPTION:
Rachialgia, whether it is cervicalgia, chest pain or low back pain, are among the most common reasons for consultation with the general practitioner in Europe.

In 2018, the therapeutic strategies for non-specific acute and subacute spine are diverse based on country clinical practice guidelines. Recommendations are rest or maintenance of normal activity, medications, surgery, psychological support, physiotherapy, acupuncture and manipulations.

Most of the guidelines, notably from Germany, Belgium, France, England and the United States, recommend spinal manipulation. In general, it can be recommended alone, or accompanied by usual care, or integrated into a multimodal treatment program. May be recommended in acute, chronic or not recommended.

The strength of osteopathy is that it tries to understand the musculoskeletal balance as a whole.

However, the differences in recommendations can be explained by the weaknesses of osteopathy, which are related to a technical and methodological problem.

The first technical problem is at the level of osteopathic clinical examination. While much of this clinical examination is based on palpatory tests, there is evidence that these range of motion palpatory tests have low sensitivity regardless of the examiner's experience.

The second methodological problem is the use of protocols.

This study attempts to propose a solution to these two problems: by proposing for the clinical examination tests of induced pain that have a greater sensitivity than palpatory tests of movements, and a comprehensive musculoskeletal treatment protocol that should allow the study to be both reliable and valid in order to be true to osteopathic values and to accept the Evidence Based Medicine methodological evaluation model.

The aim of this study is to evaluate the Osteopathic Protocol in 2 sessions (PO2).

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute or subacute cervico-dorsalgia or lumbo-dorsalgia (less than 3 months)
* Patients who gave their informed consent to participate in this study.

Exclusion Criteria:

* Patients whose specific spine is caused by inflammatory, tumor, infectious disease or back trauma in the past 3 months
* Patients with a history of back surgery and/or vertebral fracture in the past 6 months
* Patients with a motor disability related to the reason for consultation
* Pregnant women over six months.
* Patients not communicating or unable to understand the course of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline of pain level after 2 sessions | Baseline and 2 weeks
  Pain level will be collected using Visual Analog Scale (VAS) (from 0 to 10, where 10 means maximal intensity) before the first session of each protocol and one week after the second session (14 days).

SECONDARY OUTCOMES:
Percentage of pain improvement since previous visit | Week 1 and week 2
  The percent improvement will be used to assess the degree of improvement in pain experienced since the first visit.
  It will be expressed in %, the caregiver asking the patient to quantify the percentage of pain improvement on a virtual scale ranging from 0 for no improvement to 100 for complete pain disappearance.
Patient satisfaction | Week 2
  The satisfaction score will be used to assess patient satisfaction with treatment and management.
  It will be calculated on a virtual scale ranging from 0 for zero satisfaction to 10 for a total satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Michel Boeuf, Noumea, Sud, New Caledonia

IPD SHARING:
Plan to Share IPD: No